CLINICAL TRIAL: NCT00103220
Title: A Phase I Study With SJG-136 (NSC #694501) in Patients With an Advanced Solid Tumor
Brief Title: SJG-136 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01462; NCI-2012-01462 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-04076; CDR0000409581; NCI-6818; 04-076 (Other: Memorial Sloan-Kettering Cancer Center); 6818 (Other: CTEP); U01CA069856 (NIH)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 1,1'-((propane-1,3-diyl)dioxy)bis(7-methoxy-2-methylidene-1,2,3,10,11,11a-hexahydro-5H-pyrrolo(2,1-c)(1,4)benzodiazepin-5,11-dione)

ARMS (1):
- Treatment (SJG-136) (Experimental): Patients receive SJG-136 IV over 20 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: SJG-136

INTERVENTIONS:
Drug: SJG-136 — Given IV

SUMMARY:
This phase I trial is studying the side effects and best dose of SJG-136 in treating patients with advanced solid tumors. Drugs used in chemotherapy, such as SJG-136, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities, pharmacokinetic profile and the recommended phase 2 dose of SJG-136 in patients with an advanced solid tumor.

SECONDARY OBJECTIVES:

I. To determine preliminary efficacy data and evaluation of correlative markers of DNA damage and apoptosis in peripheral blood lymphocytes.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive SJG-136 intravenously (IV) over 20 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of SJG-136 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor

  * Advanced disease, defined as metastatic or unresectable disease
* Measurable indicator lesions
* Standard curative or palliative measures do not exist or are no longer effective
* Previously treated CNS metastases allowed provided patient has completed local therapy AND corticosteroids have been discontinued for at least 4 weeks
* No known leptomeningeal metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.0 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine < 1.4 mg/dL
* No congestive heart failure
* No recent myocardial infarction
* No unstable angina
* No uncontrolled hypertension
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drug
* No other significant medical history, unstable medical condition, or unstable systemic disease that would preclude study participation
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas and 8 weeks for UCN-01)
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to ≥ 25% of hematopoietic bone marrow
* Recovered from all prior therapy
* At least 4 weeks since prior investigational anticancer drugs
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2004-11; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose of SJG-136 | Day 28
  Defined as when ≤1 out of 6 patients achieve dose-limiting toxicity (DLT) at highest dose level below the maximally administered dose.

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States